CLINICAL TRIAL: NCT02154516
Title: A Consecutive Series Pilot Study Evaluating the Safety and Effectiveness of a New Hard-on-Hard Total Hip Replacement System in Patients With Non-inflammatory Arthritis With a Standard THA Metal Ion Control Group
Brief Title: Pilot Study Evaluating the Safety and Efficacy of a New Hard-on-Hard Total Hip Replacement System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011-ODHH166
Record Dates: First submitted 2014-05-13; First posted 2014-06-03 (Estimated); Results first posted 2024-12-06 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2023-04

CONDITIONS: Arthritis, Degenerative
Keywords: total hip replacement (THR); total hip arthroplasty (THA)
MeSH Terms: conditions — Osteoarthritis | interventions — Arthroplasty, Replacement, Hip

ARMS (2):
- Control Total Hip Replacement Device (Active Comparator): Total Hip replacement surgery using control device consisting of a hard-on-soft bearing or a ceramic-on-ceramic bearing which includes:
  * R3 acetabular cup, and an uncemented SYNERGY or ANTHOLOGY femoral stem
  * OXINIUM heads on polyethylene liners or
  * Ceramic heads on ceramic liners (all uncemented components)
  Interventions: Device: ODH Hip System
- Investigational Hard-on-Hard Total Hip Replacement Device (Experimental): Total Hip replacement surgery using an experimental device consisting of a hard-on-hard bearing which includes:
  * R3 acetabular cup, and an uncemented SYNERGY or ANTHOLOGY femoral stem
  * R3 ODH acetabular cup liners (sizes 38/50, 40/52, 42/54 and 44/56 mm)
  * R3 ODH femoral heads (sizes 38, 40, 42 and 44 mm)
  * Taper sleeves Ti -6AL-4V (sizes -4, +0, +4, and +8)
  Interventions: Device: ODH Hip System

INTERVENTIONS:
Device: ODH Hip System
  Other Names: Total Hip Replacement; THR; Total Hip Arthroplasty; THA

SUMMARY:
The purpose of this study is to assess the early and long term safety and efficacy of the hard-on-hard total hip replacement system (R3 ODH-ODH utilization) in patients with non-inflammatory arthritis.

ELIGIBILITY:
Inclusion Criteria:

* At least 21 years old
* Skeletally mature
* Requires primary, unilateral total hip arthroplasty due to degenerative join disease
* Preoperative Harris Hip Score of less than or equal to 70
* Meets an acceptable preoperative medical clearance and is free or treated for conditions that would pose excessive operative risk
* Given consent to participate in the study
* Able to understand the purpose of the study, his/her role, and is available for follow-up

  10 year extension:
  * Subject has completed the 2 year primary study
  * Subject has signed an Independent Ethics Committee (IEC) approved Informed Consent Form agreeing to participate in the extension study after the nature, scope and possible consequences of the study have been explained in an understandable form
  * Subject is able to fully understand the purpose of the study, his/her role as a participant in the study, and plans to be available through ten years post-operative follow-up

Exclusion Criteria:

* Diagnosis with high risk of Total Hip Arthroplasty (THA) failure
* Requires bilateral THA
* Requires revision of a prior hip replacement
* Active infection or sepsis
* History of local hip infection
* Known metastatic or neoplastic disease
* Conditions that may interfere with THA survival or outcomes
* Need for structural bone grafts to support the implant
* Contralateral lower extremity condition
* Has other joint replacements or plans for other joint replacements within 2 years
* Systemic steroid therapy within 3 months prior to surgery
* Life expectancy less than 2 years
* Intra-articular therapy within 6 months of enrollment
* Female of child-bearing age not using contraception
* Inadequate bone stock to support the device
* Moderate to severe renal insufficiency
* Emotional or neurological condition that would pre-empt ability or willingness to participate in the study
* BMI >40
* Above the knee amputation of the contralateral or ipsilateral leg
* Known allergies to the components of the devices
* Entered into another investigational study
* Is a prisoner

  10 year extension:

  • In the opinion of the surgeon, the subject's health, safety or well-being may be compromised or harmed by continuation in the extension phase or participation may not be in the subject's best interests.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2011-11-04 (Actual); Primary Completion 2022-10-18 (Actual); Study Completion 2022-10-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Baker, Principal Investigator — Entabeni Hospital; Johannes de Beer, Principal Investigator — Zuid Afrikaans Hospital
Locations (2):
- South Africa (2):
  - Entabeni Hospital, Durban
  - Zuid Afrikaans Hospital, Pretoria

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Investigational Hard-on-Hard Total Hip Replacement Device | Control Total Hip Replacement Device
Started | 20 | 6
Completed | 16 | 4
Not Completed | 4 | 2
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Removal/revision of device | 1 | 0
Not completed — Death | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Investigational Hard-on-Hard Total Hip Replacement Device | Control Total Hip Replacement Device | Total
Number analyzed (Participants) | 20 | 6 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.2 (12.48) | 56.3 (13.25) | 51.6 (12.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 4 | 11
  Male | 13 | 2 | 15
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 18 | 6 | 24
  Indian | 2 | 0 | 2
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 27 (15.94) | 86 (16.38) | 83.8 (15.75)
Treated Hip Side [Count of Participants; unit: Participants]
  Left Only | 6 | 2 | 8
  Right Only | 14 | 4 | 18
  Both Left and Right (Bilateral) | 0 | 0 | 0
Medical History - Primary Diagnosis [Count of Participants; unit: Participants]
  Osteoarthritis | 13 | 2 | 15
  Dysplasia/DDH | 4 | 2 | 6
  Avascular necrosis | 2 | 0 | 2
  Other | 1 | 0 | 1
  Missing | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Device-Related Revisions
Description: Device related revisions reported by the number of participants with a revision required (Yes/No).
Time Frame: Postoperatively through 10 years
Population: The safety population (SAF) included all participants enrolled in the study that received the study treatment with data available at the time frame indicated.
Measure: Count of Participants; unit: Participants
Arm/Group | Investigational Hard-on-Hard Total Hip Replacement Device | Control Total Hip Replacement Device
Number analyzed (Participants) | 20 | 6
Participants
  Revision Required: Yes | 1 | 0
  Revision Required: No | 19 | 6

2. Primary Outcome: Metal Ion Concentration in Whole Blood
Description: For both investigational (i.e., Investigational Hard-on-Hard Total Hip Replacement Device) and control (i.e., Control Total Hip Replacement Device) participants, metal ion concentration in whole blood were measured for Cobalt (Co), Chromium (Cr), Nickel (Ni), Titanium (Ti), Zirconium (Zr), Niobium (Nb), Molybdenum (Mo), Vanadium (V) and Aluminum (Al) at each indicated time frame.
Time Frame: 3 months, 6 months, 1 year, 2 years, 5 years, 7 years and 10 years post-operatively.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/ml)
Arm/Group | Investigational Hard-on-Hard Total Hip Replacement Device | Control Total Hip Replacement Device
Number analyzed (Participants) | 20 | 6
nanograms per milliliter (ng/ml)
  Cobalt (Co) Concentration in Whole Blood - 3 Months: number analyzed (Participants) | 20 | 5
  Cobalt (Co) Concentration in Whole Blood - 3 Months | 0.2 (0.14) | 0.3 (0.32)
  Cobalt (Co) Concentration in Whole Blood - 6 Months: number analyzed (Participants) | 19 | 5
  Cobalt (Co) Concentration in Whole Blood - 6 Months | 0.2 (0.09) | 0.2 (0.08)
  Cobalt (Co) Concentration in Whole Blood - 1 Year: number analyzed (Participants) | 19 | 5
  Cobalt (Co) Concentration in Whole Blood - 1 Year | 0.2 (0.10) | 0.2 (0.10)
  Cobalt (Co) Concentration in Whole Blood - 2 Years: number analyzed (Participants) | 19 | 5
  Cobalt (Co) Concentration in Whole Blood - 2 Years | 0.3 (0.30) | 0.2 (0.12)
  Cobalt (Co) Concentration in Whole Blood - 5 Years: number analyzed (Participants) | 19 | 5
  Cobalt (Co) Concentration in Whole Blood - 5 Years | 0.1 (0.06) | 0.1 (0.07)
  Cobalt (Co) Concentration in Whole Blood - 7 Years: number analyzed (Participants) | 16 | 4
  Cobalt (Co) Concentration in Whole Blood - 7 Years | 0.3 (0.17) | 1.0 (1.56)
  Cobalt (Co) Concentration in Whole Blood -10 Years: number analyzed (Participants) | 13 | 3
  Cobalt (Co) Concentration in Whole Blood -10 Years | 0.3 (0.12) | 0.2 (0.06)
  Chromium (Cr) Concentration in Whole Blood - 3 Months: number analyzed (Participants) | 20 | 5
  Chromium (Cr) Concentration in Whole Blood - 3 Months | 0.5 (0.18) | 0.5 (0.16)
  Chromium (Cr) Concentration in Whole Blood - 6 Months: number analyzed (Participants) | 19 | 5
  Chromium (Cr) Concentration in Whole Blood - 6 Months | 0.4 (0.04) | 0.4 (0.01)
  Chromium (Cr) Concentration in Whole Blood - 1 Year: number analyzed (Participants) | 19 | 5
  Chromium (Cr) Concentration in Whole Blood - 1 Year | 0.4 (0.09) | 0.4 (0.07)
  Chromium (Cr) Concentration in Whole Blood - 2 Years: number analyzed (Participants) | 19 | 5
  Chromium (Cr) Concentration in Whole Blood - 2 Years | 0.7 (0.56) | 0.6 (0.25)
  Chromium (Cr) Concentration in Whole Blood - 5 Years: number analyzed (Participants) | 19 | 5
  Chromium (Cr) Concentration in Whole Blood - 5 Years | 0.6 (0.10) | 0.6 (0.26)
  Chromium (Cr) Concentration in Whole Blood - 7 Years: number analyzed (Participants) | 16 | 4
  Chromium (Cr) Concentration in Whole Blood - 7 Years | 0.6 (0.21) | 0.8 (0.51)
  Chromium (Cr) Concentration in Whole Blood - 10 Years: number analyzed (Participants) | 13 | 3
  Chromium (Cr) Concentration in Whole Blood - 10 Years | 0.6 (0.51) | 0.7 (0.38)
  Nickel (Ni) Concentration in Whole Blood - 3 Months: number analyzed (Participants) | 20 | 5
  Nickel (Ni) Concentration in Whole Blood - 3 Months | 1.2 (2.67) | 0.9 (0.59)
  Nickel (Ni) Concentration in Whole Blood - 6 Months: number analyzed (Participants) | 19 | 5
  Nickel (Ni) Concentration in Whole Blood - 6 Months | 2.3 (6.99) | 0.5 (0.00)
  Nickel (Ni) Concentration in Whole Blood - 1 Year: number analyzed (Participants) | 19 | 5
  Nickel (Ni) Concentration in Whole Blood - 1 Year | 0.6 (0.20) | 0.5 (0.05)
  Nickel (Ni) Concentration in Whole Blood - 2 Years: number analyzed (Participants) | 19 | 5
  Nickel (Ni) Concentration in Whole Blood - 2 Years | 0.9 (0.55) | 0.6 (0.12)
  Nickel (Ni) Concentration in Whole Blood - 5 Years: number analyzed (Participants) | 19 | 5
  Nickel (Ni) Concentration in Whole Blood - 5 Years | 0.6 (0.22) | 0.8 (0.57)
  Nickel (Ni) Concentration in Whole Blood - 7 Years: number analyzed (Participants) | 16 | 4
  Nickel (Ni) Concentration in Whole Blood - 7 Years | 0.9 (0.29) | 0.9 (0.85)
  Nickel (Ni) Concentration in Whole Blood - 10 Years: number analyzed (Participants) | 13 | 3
  Nickel (Ni) Concentration in Whole Blood - 10 Years | 0.7 (0.18) | 1.5 (1.16)
  Titanium (Ti) Concentration in Whole Blood - 3 Months: number analyzed (Participants) | 20 | 5
  Titanium (Ti) Concentration in Whole Blood - 3 Months | 1.5 (0.62) | 1.4 (0.63)
  Titanium (Ti) Concentration in Whole Blood - 6 Months: number analyzed (Participants) | 20 | 5
  Titanium (Ti) Concentration in Whole Blood - 6 Months | 1.5 (0.41) | 1.9 (0.91)
  Titanium (Ti) Concentration in Whole Blood - 1 Year: number analyzed (Participants) | 19 | 5
  Titanium (Ti) Concentration in Whole Blood - 1 Year | 1.7 (0.35) | 2.3 (1.10)
  Titanium (Ti) Concentration in Whole Blood - 2 Years: number analyzed (Participants) | 19 | 5
  Titanium (Ti) Concentration in Whole Blood - 2 Years | 1.5 (0.66) | 1.7 (0.28)
  Titanium (Ti) Concentration in Whole Blood - 5 Years: number analyzed (Participants) | 19 | 5
  Titanium (Ti) Concentration in Whole Blood - 5 Years | 1.8 (1.12) | 1.8 (0.30)
  Titanium (Ti) Concentration in Whole Blood - 7 Years: number analyzed (Participants) | 16 | 4
  Titanium (Ti) Concentration in Whole Blood - 7 Years | 1.7 (0.60) | 1.4 (0.75)
  Titanium (Ti) Concentration in Whole Blood - 10 Years: number analyzed (Participants) | 13 | 3
  Titanium (Ti) Concentration in Whole Blood - 10 Years | 1.3 (0.52) | 2.3 (1.89)
  Zirconium (Zr) Concentration in Whole Blood - 3 Months: number analyzed (Participants) | 20 | 5
  Zirconium (Zr) Concentration in Whole Blood - 3 Months | 0.6 (0.30) | 0.2 (0.07)
  Zirconium (Zr) Concentration in Whole Blood - 6 Months: number analyzed (Participants) | 19 | 5
  Zirconium (Zr) Concentration in Whole Blood - 6 Months | 0.4 (0.11) | 0.1 (0.03)
  Zirconium (Zr) Concentration in Whole Blood - 1 Year: number analyzed (Participants) | 19 | 5
  Zirconium (Zr) Concentration in Whole Blood - 1 Year | 0.3 (0.15) | 0.1 (0.05)
  Zirconium (Zr) Concentration in Whole Blood - 2 Years: number analyzed (Participants) | 19 | 5
  Zirconium (Zr) Concentration in Whole Blood - 2 Years | 0.5 (0.27) | 0.3 (0.33)
  Zirconium (Zr) Concentration in Whole Blood - 5 Years: number analyzed (Participants) | 19 | 5
  Zirconium (Zr) Concentration in Whole Blood - 5 Years | 0.4 (0.30) | 0.2 (0.05)
  Zirconium (Zr) Concentration in Whole Blood - 7 Years: number analyzed (Participants) | 16 | 4
  Zirconium (Zr) Concentration in Whole Blood - 7 Years | 0.8 (0.64) | 0.3 (0.16)
  Zirconium (Zr) Concentration in Whole Blood - 10 Years: number analyzed (Participants) | 13 | 3
  Zirconium (Zr) Concentration in Whole Blood - 10 Years | 0.5 (0.49) | 0.2 (0.21)
  Niobium (Nb) Concentration in Whole Blood - 3 Months: number analyzed (Participants) | 20 | 5
  Niobium (Nb) Concentration in Whole Blood - 3 Months | 0.1 (0.02) | 0.1 (0.01)
  Niobium (Nb) Concentration in Whole Blood - 6 Months: number analyzed (Participants) | 19 | 5
  Niobium (Nb) Concentration in Whole Blood - 6 Months | 0.1 (0.02) | 0.1 (0.00)
  Niobium (Nb) Concentration in Whole Blood - 1 Year: number analyzed (Participants) | 19 | 5
  Niobium (Nb) Concentration in Whole Blood - 1 Year | 0.1 (0.00) | 0.1 (0.00)
  Niobium (Nb) Concentration in Whole Blood - 2 Years: number analyzed (Participants) | 19 | 5
  Niobium (Nb) Concentration in Whole Blood - 2 Years | 0.1 (0.01) | 0.1 (0.01)
  Niobium (Nb) Concentration in Whole Blood - 5 Years: number analyzed (Participants) | 19 | 5
  Niobium (Nb) Concentration in Whole Blood - 5 Years | 0.1 (0.00) | 0.1 (0.02)
  Niobium (Nb) Concentration in Whole Blood - 7 Years: number analyzed (Participants) | 16 | 4
  Niobium (Nb) Concentration in Whole Blood - 7 Years | 0.2 (0.28) | 0.1 (0.03)
  Niobium (Nb) Concentration in Whole Blood - 10 Years: number analyzed (Participants) | 13 | 3
  Niobium (Nb) Concentration in Whole Blood - 10 Years | 0.1 (0.01) | 0.0 (0.01)
  Molybdenum (Mo) Concentration in Whole Blood - 3 Months: number analyzed (Participants) | 20 | 5
  Molybdenum (Mo) Concentration in Whole Blood - 3 Months | 1.1 (0.61) | 0.9 (0.51)
  Molybdenum (Mo) Concentration in Whole Blood - 6 Months: number analyzed (Participants) | 19 | 5
  Molybdenum (Mo) Concentration in Whole Blood - 6 Months | 0.8 (0.52) | 0.7 (0.29)
  Molybdenum (Mo) Concentration in Whole Blood - 1 Year: number analyzed (Participants) | 19 | 5
  Molybdenum (Mo) Concentration in Whole Blood - 1 Year | 0.5 (0.14) | 0.5 (0.25)
  Molybdenum (Mo) Concentration in Whole Blood - 2 Years: number analyzed (Participants) | 19 | 5
  Molybdenum (Mo) Concentration in Whole Blood - 2 Years | 0.9 (0.44) | 0.6 (0.09)
  Molybdenum (Mo) Concentration in Whole Blood - 5 Years: number analyzed (Participants) | 19 | 5
  Molybdenum (Mo) Concentration in Whole Blood - 5 Years | 0.7 (0.39) | 0.5 (0.14)
  Molybdenum (Mo) Concentration in Whole Blood - 7 Years: number analyzed (Participants) | 16 | 4
  Molybdenum (Mo) Concentration in Whole Blood - 7 Years | 1.0 (0.96) | 0.6 (0.64)
  Molybdenum (Mo) Concentration in Whole Blood - 10 Years: number analyzed (Participants) | 13 | 3
  Molybdenum (Mo) Concentration in Whole Blood - 10 Years | 0.6 (0.31) | 0.8 (0.55)
  Vanadium (V) Concentration in Whole Blood - 3 Months: number analyzed (Participants) | 20 | 5
  Vanadium (V) Concentration in Whole Blood - 3 Months | 0.1 (0.17) | 0.1 (0.00)
  Vanadium (V) Concentration in Whole Blood - 6 Months: number analyzed (Participants) | 19 | 5
  Vanadium (V) Concentration in Whole Blood - 6 Months | 0.1 (0.05) | 0.1 (0.00)
  Vanadium (V) Concentration in Whole Blood - 1 Year: number analyzed (Participants) | 19 | 5
  Vanadium (V) Concentration in Whole Blood - 1 Year | 0.1 (0.06) | 0.1 (0.00)
  Vanadium (V) Concentration in Whole Blood - 2 Years: number analyzed (Participants) | 19 | 5
  Vanadium (V) Concentration in Whole Blood - 2 Years | 0.1 (0.04) | 0.1 (0.01)
  Vanadium (V) Concentration in Whole Blood - 5 Years: number analyzed (Participants) | 19 | 5
  Vanadium (V) Concentration in Whole Blood - 5 Years | 0.3 (0.65) | 0.01 (0.03)
  Vanadium (V) Concentration in Whole Blood - 7 Years: number analyzed (Participants) | 16 | 4
  Vanadium (V) Concentration in Whole Blood - 7 Years | 0.2 (0.06) | 0.2 (0.09)
  Vanadium (V) Concentration in Whole Blood - 10 Years: number analyzed (Participants) | 13 | 3
  Vanadium (V) Concentration in Whole Blood - 10 Years | 0.1 (0.14) | 0.3 (0.19)
  Aluminum (Al) Concentration in Whole Blood - 3 Months: number analyzed (Participants) | 20 | 5
  Aluminum (Al) Concentration in Whole Blood - 3 Months | 5.8 (1.61) | 5.9 (1.96)
  Aluminum (Al) Concentration in Whole Blood - 6 Months: number analyzed (Participants) | 19 | 5
  Aluminum (Al) Concentration in Whole Blood - 6 Months | 7.0 (3.80) | 6.1 (0.98)
  Aluminum (Al) Concentration in Whole Blood - 1 Year: number analyzed (Participants) | 19 | 5
  Aluminum (Al) Concentration in Whole Blood - 1 Year | 8.5 (4.62) | 10.3 (5.01)
  Aluminum (Al) Concentration in Whole Blood - 2 Years: number analyzed (Participants) | 19 | 5
  Aluminum (Al) Concentration in Whole Blood - 2 Years | 11.2 (6.86) | 7.2 (2.07)
  Aluminum (Al) Concentration in Whole Blood - 5 Years: number analyzed (Participants) | 19 | 5
  Aluminum (Al) Concentration in Whole Blood - 5 Years | 10.4 (7.20) | 9.4 (9.93)
  Aluminum (Al) Concentration in Whole Blood - 7 Years: number analyzed (Participants) | 16 | 4
  Aluminum (Al) Concentration in Whole Blood - 7 Years | 15.0 (10.50) | 10.0 (5.98)
  Aluminum (Al) Concentration in Whole Blood - 10 Years: number analyzed (Participants) | 13 | 3
  Aluminum (Al) Concentration in Whole Blood - 10 Years | 11.0 (7.02) | 7.1 (1.32)

3. Secondary Outcome: Harris Hip Score (HHS) - Investigational Hard-on-Hard Total Hip Replacement Device Only
Description: The Harris Hip Score (HHS), which ranges from 0 (worst) to 100 (best), considers information on pain, function, and range of motion. HHS was measured for Investigational Hard-on-Hard Total Hip Replacement Device only.
Time Frame: Preoperatively, 3 months, 6 months, 1 year, 2 years, 5 years, 7 years and 10 years post-operatively.
Population: The Intent to Treat (ITT) population included participants enrolled in the study with data available at the time frame indicated. The ITT did not include those that only provided retrospective data, therefore only data for the Investigational Hard-on-Hard Total Hip Replacement Device group was collected.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Investigational Hard-on-Hard Total Hip Replacement Device
Number analyzed (Participants) | 20
score on a scale
  Preoperative | 51.0 (9.48)
  3 Months | 85.6 (11.28)
  6 Months: number analyzed (Participants) | 19
  6 Months | 92.6 (9.77)
  1 Year: number analyzed (Participants) | 19
  1 Year | 94.7 (9.79)
  2 Years: number analyzed (Participants) | 19
  2 Years | 95.2 (10.21)
  5 Years: number analyzed (Participants) | 18
  5 Years | 92.9 (14.44)
  7 Years: number analyzed (Participants) | 16
  7 Years | 94.9 (12.60)
  10 Years: number analyzed (Participants) | 14
  10 Years | 97.1 (9.35)

4. Secondary Outcome: Hip Disability and Osteoarthritis Outcome Scores (HOOS)
Description: The Hip Disability and Osteoarthritis Outcome Scores (HOOS) was measured for Investigational Hard-on-Hard Total Hip Replacement Device only and included 40 items with five responses from five subcategories of Pain, Symptoms and Stiffness, Activities of Daily Living, Function in Sports and Recreational Activities, and Quality of Life to produce a total HOOS. The total HOOS scale ranged from 0 to 100, with 0 indicating the worst possible score and 100 indicating the best possible score.
Time Frame: Preoperatively, 3 months, 6 months, 1 year, 2 years, 5 years, 7 years, 10 years
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Investigational Hard-on-Hard Total Hip Replacement Device
Number analyzed (Participants) | 20
score on a scale
  Preoperative | 44.9 (19.86)
  3 Months | 83.8 (18.84)
  6 Months: number analyzed (Participants) | 19
  6 Months | 85.8 (21.08)
  1 Year: number analyzed (Participants) | 19
  1 Year | 91.8 (14.53)
  2 Years: number analyzed (Participants) | 19
  2 Years | 92.9 (14.07)
  5 Years: number analyzed (Participants) | 18
  5 Years | 85.6 (26.91)
  7 Years: number analyzed (Participants) | 17
  7 Years | 88.8 (22.95)
  10 Years: number analyzed (Participants) | 16
  10 Years | 88.4 (22.87)

5. Secondary Outcome: Radiographic Measures: Radiolucencies
Description: Radiolucencies determined by number of participants with occurrence of radiolucent lines and osteolysis (Yes/No)
Time Frame: 3 months, 6 months, 1 year, 2 years, 5 years, 7 years and 10 years post-operative
Population: The safety population (SAF) included all participants enrolled in the study that received the study treatment with data available at the time frame indicated. Data was not collected for the control total hip replacement device group at 3 months, 6 months, 1 year, and 2 years.
Measure: Count of Participants; unit: Participants
Arm/Group | Investigational Hard-on-Hard Total Hip Replacement Device | Control Total Hip Replacement Device
Number analyzed (Participants) | 20 | 5
Participants
  Radiolucent Line - 3 months: number analyzed (Participants) | 20 | 0
  Radiolucent Line - 3 months: No | 17 | 0
  Radiolucent Line - 3 months: Yes | 3 | 0
  Osteolysis - 3 months: number analyzed (Participants) | 20 | 0
  Osteolysis - 3 months: No | 17 | 0
  Osteolysis - 3 months: Yes | 3 | 0
  Radiolucent Line - 6 months: number analyzed (Participants) | 19 | 0
  Radiolucent Line - 6 months: No | 19 | 0
  Radiolucent Line - 6 months: Yes | 0 | 0
  Osteolysis - 6 months: number analyzed (Participants) | 19 | 0
  Osteolysis - 6 months: No | 18 | 0
  Osteolysis - 6 months: Yes | 1 | 0
  Radiolucent Line - 1 Year: number analyzed (Participants) | 19 | 0
  Radiolucent Line - 1 Year: No | 15 | 0
  Radiolucent Line - 1 Year: Yes | 4 | 0
  Osteolysis - 1 Year: number analyzed (Participants) | 19 | 0
  Osteolysis - 1 Year: No | 13 | 0
  Osteolysis - 1 Year: Yes | 6 | 0
  Radiolucent Line - 2 Years: number analyzed (Participants) | 19 | 0
  Radiolucent Line - 2 Years: No | 17 | 0
  Radiolucent Line - 2 Years: Yes | 2 | 0
  Osteolysis - 2 Years: number analyzed (Participants) | 19 | 0
  Osteolysis - 2 Years: No | 17 | 0
  Osteolysis - 2 Years: Yes | 2 | 0
  Radiolucent Line - 5 Years: number analyzed (Participants) | 18 | 5
  Radiolucent Line - 5 Years: No | 18 | 5
  Radiolucent Line - 5 Years: Yes | 0 | 0
  Osteolysis - 5 Years: number analyzed (Participants) | 18 | 5
  Osteolysis - 5 Years: No | 18 | 5
  Osteolysis - 5 Years: Yes | 0 | 0
  Radiolucent Line - 7 Years: number analyzed (Participants) | 17 | 4
  Radiolucent Line - 7 Years: No | 16 | 4
  Radiolucent Line - 7 Years: Yes | 1 | 0
  Osteolysis - 7 Years: number analyzed (Participants) | 17 | 4
  Osteolysis - 7 Years: No | 16 | 4
  Osteolysis - 7 Years: Yes | 1 | 0
  Radiolucent Line - 10 Years: number analyzed (Participants) | 14 | 4
  Radiolucent Line - 10 Years: No | 14 | 4
  Radiolucent Line - 10 Years: Yes | 0 | 0
  Osteolysis - 10 Years: number analyzed (Participants) | 14 | 4
  Osteolysis - 10 Years: No | 14 | 4
  Osteolysis - 10 Years: Yes | 0 | 0

6. Secondary Outcome: Radiographic Measures: Heterotopic Ossification
Description: Occurrence of Heterotopic Ossification in participants (Yes/No)
Time Frame: 3 months, 6 months, 1 year, 2 years, 5 years, 7 years and 10 years post-operative
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Investigational Hard-on-Hard Total Hip Replacement Device | Control Total Hip Replacement Device
Number analyzed (Participants) | 20 | 5
Participants
  Heterotopic Ossification - 3 Months: number analyzed (Participants) | 20 | 0
  Heterotopic Ossification - 3 Months: No Heterotopic Ossification | 18 | 0
  Heterotopic Ossification - 3 Months: Heterotopic Ossification Grade 1 | 2 | 0
  Heterotopic Ossification - 3 Months: Heterotopic Ossification Grade 2 | 0 | 0
  Heterotopic Ossification - 3 Months: Heterotopic Ossification Grade 3 | 0 | 0
  Heterotopic Ossification - 3 Months: Heterotopic Ossification Grade 4 | 0 | 0
  Heterotopic Ossification - 6 Months: number analyzed (Participants) | 19 | 0
  Heterotopic Ossification - 6 Months: No Heterotopic Ossification | 15 | 0
  Heterotopic Ossification - 6 Months: Heterotopic Ossification Grade 1 | 3 | 0
  Heterotopic Ossification - 6 Months: Heterotopic Ossification Grade 2 | 1 | 0
  Heterotopic Ossification - 6 Months: Heterotopic Ossification Grade 3 | 0 | 0
  Heterotopic Ossification - 6 Months: Heterotopic Ossification Grade 4 | 0 | 0
  Heterotopic Ossification - 1 Year: number analyzed (Participants) | 19 | 0
  Heterotopic Ossification - 1 Year: No Heterotopic Ossification | 14 | 0
  Heterotopic Ossification - 1 Year: Heterotopic Ossification Grade 1 | 4 | 0
  Heterotopic Ossification - 1 Year: Heterotopic Ossification Grade 2 | 1 | 0
  Heterotopic Ossification - 1 Year: Heterotopic Ossification Grade 3 | 0 | 0
  Heterotopic Ossification - 1 Year: Heterotopic Ossification Grade 4 | 0 | 0
  Heterotopic Ossification - 2 Years: number analyzed (Participants) | 19 | 0
  Heterotopic Ossification - 2 Years: No Heterotopic Ossification | 18 | 0
  Heterotopic Ossification - 2 Years: Heterotopic Ossification Grade 1 | 0 | 0
  Heterotopic Ossification - 2 Years: Heterotopic Ossification Grade 2 | 1 | 0
  Heterotopic Ossification - 2 Years: Heterotopic Ossification Grade 3 | 0 | 0
  Heterotopic Ossification - 2 Years: Heterotopic Ossification Grade 4 | 0 | 0
  Heterotopic Ossification - 5 Years: number analyzed (Participants) | 18 | 5
  Heterotopic Ossification - 5 Years: No Heterotopic Ossification | 16 | 4
  Heterotopic Ossification - 5 Years: Heterotopic Ossification Grade 1 | 1 | 0
  Heterotopic Ossification - 5 Years: Heterotopic Ossification Grade 2 | 1 | 1
  Heterotopic Ossification - 5 Years: Heterotopic Ossification Grade 3 | 0 | 0
  Heterotopic Ossification - 5 Years: Heterotopic Ossification Grade 4 | 0 | 0
  Heterotopic Ossification - 7 Years: number analyzed (Participants) | 17 | 4
  Heterotopic Ossification - 7 Years: No Heterotopic Ossification | 14 | 2
  Heterotopic Ossification - 7 Years: Heterotopic Ossification Grade 1 | 2 | 2
  Heterotopic Ossification - 7 Years: Heterotopic Ossification Grade 2 | 1 | 0
  Heterotopic Ossification - 7 Years: Heterotopic Ossification Grade 3 | 0 | 0
  Heterotopic Ossification - 7 Years: Heterotopic Ossification Grade 4 | 0 | 0
  Heterotopic Ossification - 10 Years: number analyzed (Participants) | 14 | 4
  Heterotopic Ossification - 10 Years: No Heterotopic Ossification | 13 | 2
  Heterotopic Ossification - 10 Years: Heterotopic Ossification Grade 1 | 0 | 2
  Heterotopic Ossification - 10 Years: Heterotopic Ossification Grade 2 | 1 | 0
  Heterotopic Ossification - 10 Years: Heterotopic Ossification Grade 3 | 0 | 0
  Heterotopic Ossification - 10 Years: Heterotopic Ossification Grade 4 | 0 | 0

7. Secondary Outcome: Radiographic Measures: Subsidence
Description: Occurrence of Subsidence in Investigational Hard-on-Hard Total Hip Replacement Device participants (Yes/No) categorized by:
  * Acetabular Cup Subsidence
  * Stem Subsidence
  * Evidence of cortical thickening
  * Acetabular component fail
  * Femoral component fail
  * Other
Time Frame: 3 months, 6 months, 1 year, 2 years, 5 years, 7 years and 10 years post-operative
Population: The safety population (SAF) included all participants enrolled in the study that received the study treatment with data available at the time frame indicated. The safety population (SAF) included all participants enrolled in the study that received the study treatment with data available at the time frame indicated. Data was not collected for the control total hip replacement device group at 3 months, 6 months, 1 year, and 2 years.
Measure: Count of Participants; unit: Participants
Arm/Group | Investigational Hard-on-Hard Total Hip Replacement Device | Control Total Hip Replacement Device
Number analyzed (Participants) | 20 | 5
Participants
  Acetabular Cup Subsidence - 3 months: number analyzed (Participants) | 20 | 0
  Acetabular Cup Subsidence - 3 months: No | 20 | 0
  Acetabular Cup Subsidence - 3 months: Yes | 0 | 0
  Stem Subsidence - 3 months: number analyzed (Participants) | 20 | 0
  Stem Subsidence - 3 months: No | 20 | 0
  Stem Subsidence - 3 months: Yes | 0 | 0
  Evidence of cortical thickening - 3 Months: number analyzed (Participants) | 20 | 0
  Evidence of cortical thickening - 3 Months: No | 20 | 0
  Evidence of cortical thickening - 3 Months: Yes | 0 | 0
  Acetabular component fail - 3 Months: number analyzed (Participants) | 20 | 0
  Acetabular component fail - 3 Months: No | 20 | 0
  Acetabular component fail - 3 Months: Yes | 0 | 0
  Femoral component fail - 3 Months: number analyzed (Participants) | 20 | 0
  Femoral component fail - 3 Months: No | 20 | 0
  Femoral component fail - 3 Months: Yes | 0 | 0
  Other - 3 Months: number analyzed (Participants) | 20 | 0
  Other - 3 Months: No | 20 | 0
  Other - 3 Months: Yes | 0 | 0
  Acetabular Cup Subsidence - 6 months: number analyzed (Participants) | 19 | 0
  Acetabular Cup Subsidence - 6 months: No | 19 | 0
  Acetabular Cup Subsidence - 6 months: Yes | 0 | 0
  Stem Subsidence - 6 Months: number analyzed (Participants) | 19 | 0
  Stem Subsidence - 6 Months: No | 19 | 0
  Stem Subsidence - 6 Months: Yes | 0 | 0
  Evidence of cortical thickening - 6 Months: number analyzed (Participants) | 19 | 0
  Evidence of cortical thickening - 6 Months: No | 18 | 0
  Evidence of cortical thickening - 6 Months: Yes | 1 | 0
  Acetabular component fail - 6 Months: number analyzed (Participants) | 19 | 0
  Acetabular component fail - 6 Months: No | 19 | 0
  Acetabular component fail - 6 Months: Yes | 0 | 0
  Femoral component fail - 6 Months: number analyzed (Participants) | 19 | 0
  Femoral component fail - 6 Months: No | 19 | 0
  Femoral component fail - 6 Months: Yes | 0 | 0
  Other- 6 Months: number analyzed (Participants) | 19 | 0
  Other- 6 Months: No | 19 | 0
  Other- 6 Months: Yes | 0 | 0
  Acetabular Cup Subsidence - 1 Year: number analyzed (Participants) | 19 | 0
  Acetabular Cup Subsidence - 1 Year: No | 19 | 0
  Acetabular Cup Subsidence - 1 Year: Yes | 0 | 0
  Stem Subsidence - 1 Year: number analyzed (Participants) | 19 | 0
  Stem Subsidence - 1 Year: No | 19 | 0
  Stem Subsidence - 1 Year: Yes | 0 | 0
  Evidence of cortical thickening - 1 Year: number analyzed (Participants) | 19 | 0
  Evidence of cortical thickening - 1 Year: No | 19 | 0
  Evidence of cortical thickening - 1 Year: Yes | 0 | 0
  Acetabular component fail - 1 Year: number analyzed (Participants) | 19 | 0
  Acetabular component fail - 1 Year: No | 19 | 0
  Acetabular component fail - 1 Year: Yes | 0 | 0
  Femoral component fail - 1 Year: number analyzed (Participants) | 19 | 0
  Femoral component fail - 1 Year: No | 19 | 0
  Femoral component fail - 1 Year: Yes | 0 | 0
  Other - 1 Year: number analyzed (Participants) | 19 | 0
  Other - 1 Year: No | 19 | 0
  Other - 1 Year: Yes | 0 | 0
  Acetabular Cup Subsidence - 2 Years: number analyzed (Participants) | 19 | 0
  Acetabular Cup Subsidence - 2 Years: No | 19 | 0
  Acetabular Cup Subsidence - 2 Years: Yes | 0 | 0
  Stem Subsidence 2 Years: number analyzed (Participants) | 19 | 0
  Stem Subsidence 2 Years: No | 19 | 0
  Stem Subsidence 2 Years: Yes | 0 | 0
  Evidence of cortical thickening - 2 Years: number analyzed (Participants) | 19 | 0
  Evidence of cortical thickening - 2 Years: No | 19 | 0
  Evidence of cortical thickening - 2 Years: Yes | 0 | 0
  Acetabular component fail - 2 Years: number analyzed (Participants) | 19 | 0
  Acetabular component fail - 2 Years: No | 19 | 0
  Acetabular component fail - 2 Years: Yes | 0 | 0
  Femoral component fail - 2 Years: number analyzed (Participants) | 19 | 0
  Femoral component fail - 2 Years: No | 19 | 0
  Femoral component fail - 2 Years: Yes | 0 | 0
  Other - 2 Years: number analyzed (Participants) | 19 | 0
  Other - 2 Years: No | 18 | 0
  Other - 2 Years: Yes | 1 | 0
  Acetabular Cup Subsidence - 5 Years: number analyzed (Participants) | 18 | 5
  Acetabular Cup Subsidence - 5 Years: No | 18 | 5
  Acetabular Cup Subsidence - 5 Years: Yes | 0 | 0
  Stem Subsidence - 5 Years: number analyzed (Participants) | 18 | 5
  Stem Subsidence - 5 Years: No | 17 | 5
  Stem Subsidence - 5 Years: Yes | 1 | 0
  Evidence of cortical thickening - 5 Years: number analyzed (Participants) | 18 | 5
  Evidence of cortical thickening - 5 Years: No | 18 | 4
  Evidence of cortical thickening - 5 Years: Yes | 0 | 1
  Acetabular component fail - 5 Years: number analyzed (Participants) | 18 | 5
  Acetabular component fail - 5 Years: No | 18 | 5
  Acetabular component fail - 5 Years: Yes | 0 | 0
  Femoral component fail - 5 Years: number analyzed (Participants) | 18 | 5
  Femoral component fail - 5 Years: No | 18 | 5
  Femoral component fail - 5 Years: Yes | 0 | 0
  Other - 5 Years: number analyzed (Participants) | 18 | 5
  Other - 5 Years: No | 17 | 5
  Other - 5 Years: Yes | 1 | 0
  Acetabular Cup Subsidence - 7 Years: number analyzed (Participants) | 17 | 4
  Acetabular Cup Subsidence - 7 Years: No | 17 | 4
  Acetabular Cup Subsidence - 7 Years: Yes | 0 | 0
  Stem Subsidence - 7 Years: number analyzed (Participants) | 17 | 4
  Stem Subsidence - 7 Years: No | 17 | 4
  Stem Subsidence - 7 Years: Yes | 0 | 0
  Evidence of cortical thickening - 7 Years: number analyzed (Participants) | 17 | 4
  Evidence of cortical thickening - 7 Years: No | 16 | 4
  Evidence of cortical thickening - 7 Years: Yes | 1 | 0
  Acetabular component fail - 7 Years: number analyzed (Participants) | 17 | 4
  Acetabular component fail - 7 Years: No | 17 | 4
  Acetabular component fail - 7 Years: Yes | 0 | 0
  Femoral component fail - 7 Years: number analyzed (Participants) | 17 | 4
  Femoral component fail - 7 Years: No | 17 | 4
  Femoral component fail - 7 Years: Yes | 0 | 0
  Other - 7 Years: number analyzed (Participants) | 17 | 4
  Other - 7 Years: No | 17 | 4
  Other - 7 Years: Yes | 0 | 0
  Acetabular Cup Subsidence - 10 Years: number analyzed (Participants) | 14 | 4
  Acetabular Cup Subsidence - 10 Years: No | 14 | 4
  Acetabular Cup Subsidence - 10 Years: Yes | 0 | 0
  Stem Subsidence - 10 Years: number analyzed (Participants) | 14 | 4
  Stem Subsidence - 10 Years: No | 14 | 4
  Stem Subsidence - 10 Years: Yes | 0 | 0
  Evidence of cortical thickening - 10 Years: number analyzed (Participants) | 14 | 4
  Evidence of cortical thickening - 10 Years: No | 13 | 4
  Evidence of cortical thickening - 10 Years: Yes | 1 | 0
  Acetabular component fail - 10 Years: number analyzed (Participants) | 14 | 4
  Acetabular component fail - 10 Years: No | 14 | 4
  Acetabular component fail - 10 Years: Yes | 0 | 0
  Femoral component fail - 10 Years: number analyzed (Participants) | 14 | 4
  Femoral component fail - 10 Years: No | 14 | 4
  Femoral component fail - 10 Years: Yes | 0 | 0
  Other - 10 Years: number analyzed (Participants) | 14 | 4
  Other - 10 Years: No | 14 | 4
  Other - 10 Years: Yes | 0 | 0

8. Secondary Outcome: Health Economic Outcomes: Surgical Blood Loss
Description: Blood loss during surgery measured in milliliters (ml) of blood
Time Frame: Intra-operative, up to 50 minutes
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milliliters (mL)
Arm/Group | Investigational Hard-on-Hard Total Hip Replacement Device | Control Total Hip Replacement Device
Number analyzed (Participants) | 20 | 6
milliliters (mL) | 324 (218.6) | 365 (164.2)

9. Secondary Outcome: Health Economic Outcomes: Length of Hospital Stay
Description: Length of stay measured by number of days spent in hospital
Time Frame: Hospital admission to discharge
Population: Length of hospital stay data was not collected as part of the 10 year extension study.
Groups:
- Investigational Hard-on-Hard Total Hip Replacement Device: Total Hip replacement surgery using an experimental device consisting of a hard-on-hard bearing which includes:
  * R3 acetabular cup, and an uncemented SYNERGY or ANTHOLOGY femoral stem
  * R3 ODH acetabular cup liners (sizes 38/50, 40/52, 42/54 and 44/56 mm)
  * R3 ODH femoral heads (sizes 38, 40, 42 and 44 mm)
  * Taper sleeves Ti -6AL-4V (sizes -4, +0, +4, and +8)
  ODH Hip System
- Control Total Hip Replacement Device: Total Hip replacement surgery using control device consisting of a hard-on-soft bearing or a ceramic-on-ceramic bearing which includes:
  * R3 acetabular cup, and an uncemented SYNERGY or ANTHOLOGY femoral stem
  * OXINIUM heads on polyethylene liners or
  * Ceramic heads on ceramic liners (all uncemented components)
  ODH Hip System
Arm/Group | Investigational Hard-on-Hard Total Hip Replacement Device | Control Total Hip Replacement Device
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Health Economic Outcomes: Operative Time
Description: Operative time in minutes from first incision into skin to time when last suture is applied for the Investigational Hard-on-Hard Total Hip Replacement Device group only
Time Frame: Intra-operative
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Investigational Hard-on-Hard Total Hip Replacement Device
Number analyzed (Participants) | 20
Minutes | 50.0 (14.9)

11. Secondary Outcome: Health Economic Outcomes: Re-Hospitalizations
Description: Re-hospitalizations measured by the number of re-admissions to hospital
Time Frame: Up to 10 years
Population: Re-hospitalizations data was not collected as part of the 10 year extension study.
Arm/Group | Investigational Hard-on-Hard Total Hip Replacement Device | Control Total Hip Replacement Device
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Surgery to 10-years
Arm/Group | Investigational Hard-on-Hard Total Hip Replacement Device | Control Total Hip Replacement Device
All-Cause Mortality (participants affected / at risk) | 2/20 | 1/6
Serious Adverse Events (participants affected / at risk) | 9/20 | 3/6
Other Adverse Events (participants affected / at risk) | 20/20 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Investigational Hard-on-Hard Total Hip Replacement Device (N=20) | Control Total Hip Replacement Device (N=6)
Kidney Stones (Renal and urinary disorders) | 1 (1) | 0 (0)
Uncontrolled Hypertension (Cardiac disorders) | 1 (1) | 0 (0)
Death from unknown cause (General disorders) | 1 (1) | 0 (0) — Death from unknown cause
Contralateral hip replacement (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
left shoulder Rotator cuff tear (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Irritable Bowel Syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0)
Depression and psychosomatic disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Gastroscopy and biopsy (Gastrointestinal disorders) | 1 (1) | 0 (0)
Worsening of prior muscle spasm and pain in study hip (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Death (General disorders) | 1 (1) | 0 (0) — Death by suicide
Bilateral inguinal hernia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Anterior right hip dislocation (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis left ankle (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis effusion left knee (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Right shoulder rotator cuff tear (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Loosening of implant stem (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Serious Adverse Device event
Fall onto right hip (replacement hip) (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Breast augmentation surgery (Surgical and medical procedures) | 1 (1) | 0 (0)
Surgery left foot (Surgical and medical procedures) | 1 (1) | 0 (0)
Sacroilliac joint pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Sacroilliac joint pain treatment (Surgical and medical procedures) | 1 (1) | 0 (0)
Haemorrhoids resulting in surgery (Vascular disorders) | 1 (1) | 0 (0)
Death (Cardiac disorders) | 0 (0) | 1 (1) — Death due to atrial fibrillation and aorta collapse
Hysterectomy (Reproductive system and breast disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Investigational Hard-on-Hard Total Hip Replacement Device (N=20) | Control Total Hip Replacement Device (N=6)
Increased Vanadium Levels (Blood and lymphatic system disorders) | 4 (4) | 2 (2)
Increased Nickel Levels (Blood and lymphatic system disorders) | 12 (12) | 4 (4)
Increased Titanium Levels (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Increased Cobalt Levels (Blood and lymphatic system disorders) | 11 (11) | 2 (2)
Increased Chromium Levels (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Increased Niobium Levels (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
Rash at operative site (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Greater trochanter bursitis R hip (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Hypertension (Cardiac disorders) | 5 (5) | 1 (1)
Intermittent back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis left hip (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Pain and noise in right hip (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Benign prostate hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Hypotension (Cardiac disorders) | 1 (1) | 0 (0)
Rash on back (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Gout (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Hip noise (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0)
Fall (Musculoskeletal and connective tissue disorders) | 1 (3) | 0 (0) — Subject works on farm - injury prone
Chest pain and shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Right knee pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Femoral nerve impingement right leg (Nervous system disorders) | 1 (1) | 0 (0)
Low oxygen levels (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sacroilliac pain (Musculoskeletal and connective tissue disorders) | 1 (3) | 0 (0)
Left tennis elbow (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Surgery-left foot (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Diabetes - new (Endocrine disorders) | 1 (1) | 0 (0)
Polyuria and hematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Vomitting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Kidney stones (Renal and urinary disorders) | 1 (1) | 0 (0)
Pain in operative hip (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Muscle spasm (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rash - jugular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Peripheral neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Urinary Tract Infection (Renal and urinary disorders) | 1 (1) | 0 (0)
Surgical site reaction (Infections and infestations) | 1 (1) | 0 (0)
Perineal nerve weakness left foot (Nervous system disorders) | 1 (1) | 0 (0)
rash - left foot (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Swelling below left fibular head (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Urine retention after catheter removal (Renal and urinary disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastroscopy (Gastrointestinal disorders) | 1 (1) | 0 (0)
Muscle spasm (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) — location not specified
Severe depression (Psychiatric disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Urine retention - unknown cause (Renal and urinary disorders) | 1 (1) | 0 (0)
Trochanter bursitis left hip (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Fall on operative hip (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rash on upper right arm (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Fall on contralateral hip (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
This study was initially conducted as a pilot study to assess early safety of the ODH on ODH Total Hip System in a small group of participants for up to two years. The study was then extended to include safety data for up to ten years. Imbalance of study arms and small sample size limits the amount of statistical conclusions the study can make. Not all data for Control participants were collected in every outcome measure, limiting the ability to compare the two arms.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2017-01-19): https://cdn.clinicaltrials.gov/large-docs/16/NCT02154516/Prot_000.pdf
  • Statistical Analysis Plan (2018-11-26): https://cdn.clinicaltrials.gov/large-docs/16/NCT02154516/SAP_001.pdf